CLINICAL TRIAL: NCT05707351
Title: A Phase 3, Prospective, Multicenter, Open-label Study of Efficacy, Safety, and Pharmacokinetics of PEGylated Recombinant Factor VIII (ADYNOVATE) Administered for Prophylaxis and Treatment of Bleeding in Chinese Previously Treated Patients With Severe Hemophilia A (FVIII <1%)
Brief Title: A Study of Adynovate in Previously Treated Chinese Teenagers and Adults With Severe Hemophilia A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-660-3001; 2023-000502-26 (EudraCT Number)
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — BAX 855; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adynovate 45±5 IU/kg (Experimental): Participants received prophylactic treatment with Adynovate (45 [±5] IU/kg), infusion, IV, twice weekly, for at least 50 EDs, or approximately 28 weeks.
  Interventions: Biological: Adynovate

INTERVENTIONS:
Biological: Adynovate — Adynovate was injected intravenously using an appropriately sized syringe as a bolus infusion over a period of less than or equal to (<=) 5 minutes (maximum infusion rate, 10 milliliters per minute [mL/min]).
  Other Names: Antihemophilic Factor (recombinant) PEGylated, Rurioctocog Alfa Pegol

SUMMARY:
The main aim of the study is to determine how well Adynovate works to decrease bleeding in previously treated Chinese men and boys with severe hemophilia A when given prophylactically.

Participants will be treated with Adynovate twice a week for 26 weeks or until participants have received 50 days of treatment with Adynovate (whichever takes longer). Participants will need to visit their study clinic several times during their participation.

ELIGIBILITY:
Inclusion Criteria:

1. Participant and/or legally authorized representative must voluntarily sign a written informed consent form (ICF) after all relevant aspects of the study have been explained and discussed with the Participant. For the participants less than (<) 18 years old, participants will give assent AND their parents/legally authorized representative should sign the ICF accordingly.
2. Participant and/or legally authorized representative understands and is willing and able to comply with all requirements of the study protocol.
3. Participant should be ethnic Chinese.
4. Participant is 12 to 65 years of age at screening and male.
5. Participant has severe hemophilia A (FVIII clotting activity <1 percent [%]) as confirmed by the central laboratory at screening after a washout period of at least 72 to 96 hours.
6. The last on-demand or prophylactic treatment received is within 3 months before screening.
7. Participant has documented previous treatment with plasma-derived FVIII concentrates or recombinant FVIII for greater than (>) 150 EDs.
8. Participant is human immunodeficiency virus (HIV)-negative, or HIV-positive with stable disease and CD4+ count greater than or equal to (>=) 200 cells per cubic millimeter (/mm^3).
9. Participant is hepatitis C virus (HCV) negative by antibody testing (if positive, additional polymerase chain reaction testing will be performed to confirm), as confirmed at screening; or HCV-positive with chronic stable hepatitis, as assessed by the investigator.

Exclusion Criteria:

1. Participant has detectable FVIII inhibitory antibodies (>=0.6 Bethesda units [BU] per milliliter [/mL] using the Nijmegen modification of the Bethesda assay) as confirmed by the central laboratory at screening.
2. Participant has a confirmed history of FVIII inhibitory antibodies (>=0.6 BU using the Nijmegen modification of the Bethesda assay or >=0.6 BU using the Bethesda assay) at any time prior to screening.
3. Participant has a known hypersensitivity to Adynovate or ADVATE or any of the components of the study drugs, such as mouse or hamster proteins, or other FVIII products.
4. Participant has been diagnosed with an inherited or acquired hemostatic defect other than hemophilia A (example, qualitative platelet defect or von Willebrand's disease).
5. Participant has severe hepatic dysfunction (example, >=5 times the upper limit of normal [ULN] for alanine aminotransferase [ALT] or aspartate aminotransferase [AST], a recent or persistent international normalized ratio [INR] >1.5, as confirmed by the local laboratory at screening).
6. Participant has severe renal impairment (serum creatinine >1.5 times the ULN) as confirmed by the local laboratory at screening.
7. Participant is planned or likely to undergo major surgery during the study period.
8. Participant has current or recent (<30 days) use of other PEGylated drugs before study participation or scheduled use of such drugs during study participation.
9. Participant has received emicizumab therapy within 6 months of screening.
10. Participant is currently receiving, or scheduled to receive during the study, an immunomodulating drug (example, systemic corticosteroid agent at a dose equivalent to hydrocortisone >10 milligram per day [mg/day], or alpha-interferon) other than antiretroviral chemotherapy.
11. Participant has participated in another clinical study involving the use of an investigational product (IP) other than Adynovate or an investigational device within 30 days before the screening visit or is scheduled to participate in another clinical study involving an IP or investigational device during this study.
12. Participant has a medical, psychiatric, or cognitive illness or recreational drug/alcohol use that, in the opinion of the investigator, would affect participant safety or compliance.
13. Participant, in the opinion of the investigator, is unable or unwilling to comply with the study protocol.

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (12):
- China (12):
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing
  - Xiangya Hospital of Central South University, Changsha
  - Fujian Medical University Union Hospital, Fuzhou
  - Nanfang Hospital Southern Medical University, Guangzhou
  - Anhui Province Hospital, Hefei
  - Jinan Central Hospital, Jinan
  - Shenzhen Second People's Hospital, Shenzhen
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/46da5667215042fa?idFilter=%5B%22TAK-660-3001%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at various investigative sites in China from 27 March 2023 to 05 September 2024.
Pre-assignment Details: Participants with a diagnosis of severe hemophilia A were enrolled in this study to receive Adynovate (45 [±5] international units per kilogram [IU/kg]), infusion, intravenously (IV).
Groups:
- Adynovate: Participants received prophylactic treatment with Adynovate (45 [±5] IU/kg), infusion, IV, twice weekly, for at least 50 exposure days (EDs), or approximately 28 weeks.
Period: Overall Study
Arm/Group | Adynovate
Started | 37
Completed | 34
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Reason Not Specified | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all participants who were assigned to receive a treatment regimen of Adynovate.
Groups:
- Adynovate: Participants received prophylactic treatment with Adynovate (45 [±5] IU/kg), infusion, IV, twice weekly, for at least 50 EDs, or approximately 28 weeks.
Arm/Group | Adynovate
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.1 (8.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 37
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Annualized Bleeding Rates (ABR)
Description: Total ABR was defined as the number of treated and non-treated bleeding episodes (BEs) that occurred during the treatment period, calculated as, ABR= number of unique bleeds during treatment period/(length of treatment period [days]/365.25). Total ABR for all BEs, spontaneous or traumatic, recorded in the participant's electronic diary and/or recorded in the physician/nurse/study site notes were reported.
Time Frame: Baseline through study completion or ≥50 EDs whichever occurred last (approximately 28 weeks)
Population: The FAS included all participants who were assigned to receive a treatment regimen of Adynovate.
Measure: Mean (Standard Deviation); unit: bleeds per year
Arm/Group | Adynovate
Number analyzed (Participants) | 37
bleeds per year | 4.1 (13.61)

2. Secondary Outcome: ABR Based on Bleeding Site
Description: ABR= number of unique bleeds during treatment period/(length of treatment period [days]/365.25). ABR for BEs based on bleeding site: joint or non-joint, recorded in the participant's electronic diary and/or recorded in the physician/nurse/study site notes were reported.
Time Frame: Baseline through study completion or ≥50 EDs whichever occurred last (approximately 28 weeks)
Population: The FAS included all participants who were assigned to receive a treatment regimen of Adynovate.
Measure: Mean (Standard Deviation); unit: bleeds per year
Arm/Group | Adynovate
Number analyzed (Participants) | 37
bleeds per year
  Bleeding Site: Joint | 2.7 (8.35)
  Bleeding Site: Non-Joint | 1.4 (5.48)

3. Secondary Outcome: ABR Based on Bleeding Cause
Description: ABR= number of unique bleeds during treatment period/(length of treatment period [days]/365.25). ABR for BEs based on bleeding cause: spontaneous/unknown or injury, recorded in the participant's electronic diary and/or recorded in the physician/nurse/study site notes were reported.
Time Frame: Baseline through study completion or ≥50 EDs whichever occurred last (approximately 28 weeks)
Population: The FAS included all participants who were assigned to receive a treatment regimen of Adynovate.
Measure: Mean (Standard Deviation); unit: bleeds per year
Arm/Group | Adynovate
Number analyzed (Participants) | 37
bleeds per year
  Bleeding Cause: Spontaneous/Unknown | 3.8 (13.65)
  Bleeding Cause: Injury | 0.3 (0.99)

4. Secondary Outcome: Number of Adynovate Infusions Per Week During the Prophylactic Treatment Period
Time Frame: Baseline through study completion or ≥50 EDs whichever occurred last (approximately 28 weeks)
Population: The FAS included all participants who were assigned to receive a treatment regimen of Adynovate.
Measure: Mean (Standard Deviation); unit: infusions per week
Arm/Group | Adynovate
Number analyzed (Participants) | 37
infusions per week | 2.003 (0.0563)

5. Secondary Outcome: Number of Adynovate Infusions Per Month During the Prophylactic Treatment Period
Time Frame: Baseline through study completion or ≥50 EDs whichever occurred last (approximately 28 weeks)
Population: The FAS included all participants who were assigned to receive a treatment regimen of Adynovate.
Measure: Mean (Standard Deviation); unit: infusions per month
Arm/Group | Adynovate
Number analyzed (Participants) | 37
infusions per month | 8.711 (0.2447)

6. Secondary Outcome: Weight-adjusted Consumption of Adynovate Per Week During the Prophylactic Treatment Period
Description: Weight-adjusted consumption (IU/kg) was derived as the total units infused (IU) divided by the last available body weight (kg) prior to the infusion.
Time Frame: Baseline through study completion or ≥50 EDs whichever occurred last (approximately 28 weeks)
Population: The FAS included all participants who were assigned to receive a treatment regimen of Adynovate.
Measure: Mean (Standard Deviation); unit: IU/kg per week
Arm/Group | Adynovate
Number analyzed (Participants) | 37
IU/kg per week | 89.637 (3.6807)

7. Secondary Outcome: Weight-adjusted Consumption of Adynovate Per Month During the Prophylactic Treatment Period
Description: as for outcome 6
Time Frame: Baseline through study completion or ≥50 EDs whichever occurred last (approximately 28 weeks)
Population: The FAS included all participants who were assigned to receive a treatment regimen of Adynovate.
Measure: Mean (Standard Deviation); unit: IU/kg per month
Arm/Group | Adynovate
Number analyzed (Participants) | 37
IU/kg per month | 389.760 (16.0045)

8. Secondary Outcome: Percentage of Participants With Zero Bleeding Episodes During the Study
Description: Percentages were rounded off to the nearest single decimal place.
Time Frame: Baseline through study completion or ≥50 EDs whichever occurred last (approximately 28 weeks)
Population: The FAS included all participants who were assigned to receive a treatment regimen of Adynovate.
Measure: Number; unit: percentage of participants
Arm/Group | Adynovate
Number analyzed (Participants) | 37
percentage of participants | 54.1

9. Secondary Outcome: Average Time Interval Between Bleeding Episodes (BEs)
Description: Average time interval between bleeding episodes (days)= Length of treatment period (days)/ Number of unique bleeds during treatment period. Average time interval was computed for participants with more than 1 unique BEs.
Time Frame: Baseline through study completion or ≥50 EDs whichever occurred last (approximately 28 weeks)
Population: The FAS included all participants who were assigned to receive a treatment regimen of Adynovate. Overall number of participants analyzed is the number of participants with more than 1 unique BEs.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Adynovate
Number analyzed (Participants) | 9
days | 61.869 (30.9437)

10. Secondary Outcome: Number of Bleeding Events in Each Category of Hemostatic Efficacy Rating at Resolution of Breakthrough Bleeding Episode
Description: Hemostatic efficacy for treatment of BEs was rated on 4-point Likert scale as: excellent=full relief of pain and cessation of objective signs of bleeding after a single infusion, no additional infusion is required for the control of bleeding and administration of further infusion to maintain hemostasis would not affect the scoring; good=definite pain relief and/or improvement in signs of bleeding after a single infusion, possibly requires more than 2 infusions for complete resolution and administration of further infusion to maintain hemostasis would not affect the scoring; fair=probable and/or slight relief of pain and slight improvement in signs of bleeding after a single infusion, required multiple infusions for complete resolution; none=no improvement of signs or symptoms or conditions worsen. Missing indicates the number of unique bleeding episodes without any overall hemostatic efficacy rating at resolution of breakthrough bleeding episode.
Time Frame: Baseline through study completion or ≥50 EDs whichever occurred last (approximately 28 weeks)
Population: The FAS included all participants who were assigned to receive a treatment regimen of Adynovate. Overall number of participants analyzed is the number of participants with treated bleeding episodes.
Measure: Number; unit: bleeding events
Units Other Than Participants: bleeding episodes
Arm/Group | Adynovate
Number analyzed (Participants) | 14
Number analyzed (bleeding episodes) | 31
bleeding events
  Excellent | 7
  Good | 14
  Fair | 4
  None | 0
  Missing | 6

11. Secondary Outcome: Number of Adynovate Infusions Per Bleeding Episode
Time Frame: Baseline through study completion or ≥50 EDs whichever occurred last (approximately 28 weeks)
Population: The Safety Analysis Set (SAS) included all participants treated with at least 1 Adynovate dose. Overall number of participants analyzed is the number of participants with treated bleeding episodes.
Measure: Mean (Standard Deviation); unit: infusions/bleeding episode
Units Other Than Participants: treated bleeding episodes
Arm/Group | Adynovate
Number analyzed (Participants) | 14
Number analyzed (treated bleeding episodes) | 31
infusions/bleeding episode | 2.839 (2.9337)

12. Secondary Outcome: Weight-adjusted Consumption of Adynovate Per Bleeding Episode
Description: as for outcome 6
Time Frame: Baseline through study completion or ≥50 EDs whichever occurred last (approximately 28 weeks)
Population: The SAS included all participants treated with at least 1 Adynovate dose. Overall number of participants analyzed is the number of participants with treated bleeding episodes.
Measure: Mean (Standard Deviation); unit: IU/kg per bleeding episode
Units Other Than Participants: treated bleeding episodes
Arm/Group | Adynovate
Number analyzed (Participants) | 14
Number analyzed (treated bleeding episodes) | 31
IU/kg per bleeding episode | 77.766 (81.7538)

13. Secondary Outcome: Number of Minor Surgeries With Hemostatic Efficacy Based on Global Hemostatic Efficacy Assessment (GHEA) Score as Assessed by the Operating Surgeon/Investigator
Description: GHEA score consisted of 3 individual rating scales: (1) Intra-operative Efficacy Assessment Scale, (2) Post-operative Efficacy Assessment Scale, and (3) Peri-operative Efficacy Assessment Scale. Each rating scale is based on 4 points scale ranging from: 3 (Excellent), 2 (Good), 1 (Fair), and 0 (None). The scores of 3 individual ratings scales were added together to form a GHEA score. Total score ranged from 0 to 9, where scores evaluate as: excellent (7 to 9), good (5 to 7), fair (3 to 4), and none (0 to 2). For a GHEA score of 7 to be rated "excellent" no individual assessment scores could be less than (<) 2 and at least 1 assessment score had to be equal to (=) 3; otherwise a score of 7 was rated "good".
Time Frame: Baseline through study completion or ≥50 EDs whichever occurred last (approximately 28 weeks)
Population: The FAS included all participants treated with at least 1 Adynovate dose. Only participants with hemostatic efficacy were to be assessed for this outcome measure. Overall number analyzed is zero as there were no participants who met the hemostatic assessment criteria for this outcome measure.
Arm/Group | Adynovate
Number analyzed (Participants) | 0

14. Secondary Outcome: Volume of Actual and Predicted Intra-operative and Post-operative Blood Loss After the Surgery as Assessed by the Operating Surgeon/Investigator
Time Frame: Post-operative: Day 1 and at discharge Week 26
Population: The FAS included all participants treated with at least 1 Adynovate dose. Only participants with blood loss for minor surgeries were to be assessed for this outcome measure. Overall number of participants analyzed is zero as there were no participants with blood loss for minor surgeries.
Arm/Group | Adynovate
Number analyzed (Participants) | 0

15. Secondary Outcome: Number of Participants Who Required Perioperative Transfusion of Blood, Red Blood Cells, Platelets, and Other Blood Products
Time Frame: Baseline through study completion or ≥50 EDs whichever occurred last (approximately 28 weeks)
Population: The FAS included all participants treated with at least 1 Adynovate dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Adynovate
Number analyzed (Participants) | 37
Participants | 0

16. Secondary Outcome: Daily Intra-Operative and Post-Operative Weight-Adjusted Consumption Dose of Adynovate
Time Frame: Baseline through study completion or ≥50 EDs whichever occurred last (approximately 28 weeks)
Population: The FAS included all participants treated with at least 1 Adynovate dose. Only participants who were administered Adynovate for minor surgeries were to be assessed for this outcome measure. Overall number of participants analyzed is zero as no participants were administered Adynovate for minor surgeries.
Arm/Group | Adynovate
Number analyzed (Participants) | 0

17. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Treatment-emergent Adverse Events (Serious TEAEs)
Description: An adverse event (AE): any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to medicinal product. TEAE: any AE either reported for the first time or worsening of a pre-existing event after first dose of study drug and within 30 days of the last administration of study drug. Serious TEAEs: any untoward medical occurrence that: 1) results in death, 2) is life-threatening, 3) requires inpatient hospitalization or prolongation of existing hospitalization, 4) results in persistent or significant disability/incapacity, 5) leads to a congenital anomaly/birth defect in the offspring of the participant or 6) is a medically important.
Time Frame: Up to approximately 28 weeks
Population: The SAS included all participants treated with at least 1 Adynovate dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Adynovate
Number analyzed (Participants) | 37
Participants
  TEAEs | 16
  Serious TEAEs | 1

18. Secondary Outcome: Number of Participants With Confirmed Inhibitory Antibodies to Factor VIII (FVIII), Binding Immunoglobulin G (IgG) and Immunoglobulin M (IgM) Antibodies to Adynovate and Chinese Hamster Ovary (CHO) Protein
Time Frame: Up to approximately 28 weeks
Population: The SAS included all participants treated with at least 1 Adynovate dose. Number analyzed is the number of participants with data available for analysis for the specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Adynovate
Number analyzed (Participants) | 37
Participants
  Inhibitory Antibodies to FVIII | 0
  Binding IgG Antibodies to Adynovate: number analyzed (Participants) | 31
  Binding IgG Antibodies to Adynovate | 0
  Binding IgM Antibodies to Adynovate: number analyzed (Participants) | 31
  Binding IgM Antibodies to Adynovate | 0
  Binding Antibodies to CHO Proteins | 0

19. Secondary Outcome: FVIII Activity Level in Plasma Assessed by a 1-stage Clotting Assay
Description: As per planned analysis, data for this outcome measure was collected and reported for initial pharmacokinetic (PK) assessment and second PK assessment. The initial PK assessment was performed prior to the baseline visit at Day -1. The second PK assessment was performed during the Week 20 visit. FVIII activity level reported was corrected for pre-infusion measurement.
Time Frame: Day -1 and Week 20: pre-infusion, post-infusion at multiple time-points up to 96 hours
Population: The Pharmacokinetic Full Analysis Set (PK FAS) included all participants who consented to PK evaluation, were treated with at least 1 Adynovate dose, and had at least 1 evaluable PK concentration post dose. Number analyzed is the number of participants with data available for analysis at the specified time-point.
Measure: Mean (Standard Deviation); unit: International units per deciliter(IU/dL)
Arm/Group | Adynovate
Number analyzed (Participants) | 15
International units per deciliter(IU/dL)
  Initial PK Assessment: Pre-Infusion | 0.00 (0.000)
  Initial PK Assessment: Post-Infusion, 30 Minutes: number analyzed (Participants) | 14
  Initial PK Assessment: Post-Infusion, 30 Minutes | 112.02 (26.739)
  Initial PK Assessment: Post-Infusion: 1 Hour: number analyzed (Participants) | 14
  Initial PK Assessment: Post-Infusion: 1 Hour | 106.67 (22.066)
  Initial PK Assessment: Post-Infusion: 2 Hours | 94.64 (32.185)
  Initial PK Assessment: Post-Infusion: 4 Hours | 87.67 (21.186)
  Initial PK Assessment: Post-Infusion: 8 Hours | 71.87 (16.929)
  Initial PK Assessment: Post-Infusion: 12 Hours | 58.96 (14.378)
  Initial PK Assessment: Post-Infusion: 24 Hours | 37.24 (11.573)
  Initial PK Assessment: Post-Infusion: 48 Hours | 14.60 (7.616)
  Initial PK Assessment: Post-Infusion: 72 Hours | 5.17 (3.876)
  Initial PK Assessment: Post-Infusion: 96 Hours | 2.06 (2.040)
  Second PK Assessment: Pre-Infusion: number analyzed (Participants) | 14
  Second PK Assessment: Pre-Infusion | 0.00 (0.000)
  Second PK Assessment: Post-Infusion, 30 Minutes: number analyzed (Participants) | 13
  Second PK Assessment: Post-Infusion, 30 Minutes | 109.75 (18.192)
  Second PK Assessment: Post-Infusion: 1 Hour: number analyzed (Participants) | 14
  Second PK Assessment: Post-Infusion: 1 Hour | 109.51 (20.705)
  Second PK Assessment: Post-Infusion: 2 Hours: number analyzed (Participants) | 14
  Second PK Assessment: Post-Infusion: 2 Hours | 98.82 (20.196)
  Second PK Assessment: Post-Infusion: 4 Hours: number analyzed (Participants) | 13
  Second PK Assessment: Post-Infusion: 4 Hours | 86.41 (9.587)
  Second PK Assessment: Post-Infusion: 8 Hours: number analyzed (Participants) | 14
  Second PK Assessment: Post-Infusion: 8 Hours | 73.57 (15.750)
  Second PK Assessment: Post-Infusion: 12 Hours: number analyzed (Participants) | 13
  Second PK Assessment: Post-Infusion: 12 Hours | 62.31 (14.766)
  Second PK Assessment: Post-Infusion: 24 Hours: number analyzed (Participants) | 14
  Second PK Assessment: Post-Infusion: 24 Hours | 40.53 (11.918)
  Second PK Assessment: Post-Infusion: 48 Hours: number analyzed (Participants) | 14
  Second PK Assessment: Post-Infusion: 48 Hours | 16.13 (8.275)
  Second PK Assessment: Post-Infusion: 72 Hours: number analyzed (Participants) | 14
  Second PK Assessment: Post-Infusion: 72 Hours | 7.20 (4.754)
  Second PK Assessment: Post-Infusion: 96 Hours: number analyzed (Participants) | 13
  Second PK Assessment: Post-Infusion: 96 Hours | 3.25 (2.811)

20. Secondary Outcome: Incremental Recovery Over Time During Adynovate Prophylactic Treatment
Description: Incremental recovery (IR) was calculated as IR (international units per deciliter)/(international units per kilogram [(IU/dL)/(IU/kg)] = [PostFVIII (IU/dL)-PreFVIII (IU/dL)]/Weight Adjusted Dose (IU/kg).
Time Frame: Baseline, Week 6, and Study Completion (approximately Week 28)
Population: The SAS included all participants treated with at least 1 Adynovate dose. Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis at the specified time-point.
Measure: Mean (Standard Deviation); unit: (IU/dL)/(IU/kg)
Arm/Group | Adynovate
Number analyzed (Participants) | 34
(IU/dL)/(IU/kg)
  Baseline | 2.4777 (0.67876)
  Week 6: number analyzed (Participants) | 31
  Week 6 | 2.5147 (0.64379)
  Study Completion: number analyzed (Participants) | 31
  Study Completion | 2.4083 (0.50714)

21. Secondary Outcome: Pre-dose Level of FVIII Activity in Plasma
Time Frame: Baseline, Weeks 2, 6, 12, and Study Completion (approximately Week 28): Within 30 minutes pre-infusion
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Adynovate
Number analyzed (Participants) | 36
IU/dL
  Baseline | 0.06 (0.232)
  Week 2: number analyzed (Participants) | 29
  Week 2 | 3.28 (4.999)
  Week 6: number analyzed (Participants) | 31
  Week 6 | 2.91 (2.802)
  Week 12: number analyzed (Participants) | 31
  Week 12 | 3.61 (3.994)
  Study Completion | 7.06 (16.365)

22. Secondary Outcome: Pre-dose Level of FVIII Antigen in Plasma
Description: IU/mL stands for international units per milliliter.
Time Frame: Baseline, Weeks 2, 6, 12, 20, and Study Completion (approximately Week 28): Within 30 minutes pre-infusion
Population: The SAS included all participants treated with at least 1 Adynovate dose. Number analyzed is the number of participants with data available for analysis at the specified time-point.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Adynovate
Number analyzed (Participants) | 37
IU/mL
  Baseline | 0.0276 (0.06577)
  Week 2: number analyzed (Participants) | 36
  Week 2 | 0.0782 (0.07888)
  Week 6: number analyzed (Participants) | 35
  Week 6 | 0.0689 (0.04518)
  Week 12: number analyzed (Participants) | 34
  Week 12 | 0.0649 (0.04286)
  Week 20: number analyzed (Participants) | 14
  Week 20 | 0.0856 (0.05404)
  Study Completion | 0.1011 (0.11326)

23. Secondary Outcome: Pre-dose Level of Von Willebrand Factor (VWF) Antigen in Plasma
Time Frame: Baseline, Weeks 2, 6, 12, 20, and Study Completion (approximately Week 28): Within 30 minutes pre-infusion
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percent (%)
Arm/Group | Adynovate
Number analyzed (Participants) | 37
percent (%)
  Baseline | 83.69 (35.967)
  Week 2: number analyzed (Participants) | 36
  Week 2 | 84.46 (30.811)
  Week 6: number analyzed (Participants) | 35
  Week 6 | 84.99 (34.216)
  Week 12: number analyzed (Participants) | 34
  Week 12 | 86.57 (30.024)
  Week 20: number analyzed (Participants) | 14
  Week 20 | 91.26 (34.240)
  Study Completion | 90.26 (31.714)

24. Secondary Outcome: Clearance (CL) for FVIII Activity Following an Initial Single Dose and Steady-state Dose of Adynovate
Description: Clearance reported was calculated based on pre-infusion corrected concentration data. As per planned analysis, data for this outcome measure was collected and reported for initial PK assessment and second PK assessment. The initial PK assessment was performed prior to the baseline visit at Day -1. The second PK assessment was performed during the Week 20 visit. [(dL/h)/kg] stands for deciliters per hour per kilogram.
Time Frame: Day -1 and Week 20: pre-infusion, post-infusion at multiple timepoints up to 96 hours
Population: The Pharmacokinetic Analysis Set (PK AS), a subset of the PK FAS, included all PK participants who received at least 1 Adynovate PK dose with a sufficient number of evaluable PK concentrations post dose for the estimation of PK parameters using a noncompartmental analysis (NCA). Number analyzed is the number of participants with data available for analysis at the specified time-point.
Measure: Mean (Standard Deviation); unit: (dL/h)/kg
Arm/Group | Adynovate
Number analyzed (Participants) | 15
(dL/h)/kg
  Initial PK Assessment | 0.0206 (0.00629)
  Second PK Assessment: number analyzed (Participants) | 14
  Second PK Assessment | 0.0192 (0.00594)

25. Secondary Outcome: Volume of Distribution for FVIII Activity Following an Initial Single Dose and Steady-state Dose of Adynovate
Description: Volume of distribution was calculated based on pre-infusion corrected concentration data. As per planned analysis, data for this outcome measure was collected and reported for initial PK assessment and second PK assessment. The initial PK assessment was performed prior to the baseline visit at Day -1. The second PK assessment was performed during the Week 20 visit.
Time Frame: Day -1 and Week 20: pre-infusion, post-infusion at multiple timepoints up to 96 hours
Population: The PK AS, a subset of the PK FAS, included all PK participants who received at least 1 Adynovate PK dose with a sufficient number of evaluable PK concentrations post dose for the estimation of PK parameters using an NCA. Number analyzed is the number of participants with data available for analysis at the specified time-point.
Measure: Mean (Standard Deviation); unit: deciliters per kilogram (dL/kg)
Arm/Group | Adynovate
Number analyzed (Participants) | 15
deciliters per kilogram (dL/kg)
  Initial PK Assessment | 0.458 (0.107)
  Second PK Assessment: number analyzed (Participants) | 14
  Second PK Assessment | 0.480 (0.0953)

26. Secondary Outcome: Area Under the Concentration Versus Time Curve From 0 to 96 Hours (AUC0-96) for FVIII Activity Following an Initial Single Dose and Steady-state Dose of Adynovate
Description: AUC0-96 was calculated based on pre-infusion corrected concentration data. As per planned analysis, data for this outcome measure was collected and reported for initial PK assessment and second PK assessment. The initial PK assessment was performed prior to the baseline visit at Day -1. The second PK assessment was performed during the Week 20 visit. h*IU/dL stands for hour*international units per deciliter.
Time Frame: Day -1 and Week 20: pre-infusion, post-infusion at multiple timepoints up to 96 hours
Population: The PK AS, a subset of the PK FAS, included all PK participants who received at least 1 Adynovate PK dose with a sufficient number of evaluable PK concentrations post dose for the estimation of PK parameters using an NCA. Number analyzed is the number of participants with data available for analysis for the specified time-point.
Measure: Mean (Standard Deviation); unit: h*IU/dL
Arm/Group | Adynovate
Number analyzed (Participants) | 15
h*IU/dL
  Initial PK Assessment | 2348 (737)
  Second PK Assessment: number analyzed (Participants) | 14
  Second PK Assessment | 2582 (736)

27. Secondary Outcome: Maximum Concentration (Cmax) for FVIII Activity Following an Initial Single Dose and Steady-state Dose of Adynovate
Description: Cmax was calculated based on pre-infusion corrected concentration data. As per planned analysis, data for this outcome measure was collected and reported for initial PK assessment and second PK assessment. The initial PK assessment was performed prior to the baseline visit at Day -1. The second PK assessment was performed during the Week 20 visit.
Time Frame: Day -1 and Week 20: pre-infusion, post-infusion at multiple timepoints up to 96 hours
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Adynovate
Number analyzed (Participants) | 15
IU/dL
  Initial PK Assessment | 113 (26.1)
  Second PK Assessment: number analyzed (Participants) | 14
  Second PK Assessment | 115 (20.0)

28. Secondary Outcome: Pre-dose Concentration (Cpredose) for FVIII Activity Following an Initial Single Dose and Steady-state Dose of Adynovate
Description: Cpredose was calculated based on pre-infusion corrected concentration data. As per planned analysis, data for this outcome measure was collected and reported for initial PK assessment and second PK assessment. The initial PK assessment was performed prior to the baseline visit at Day -1. The second PK assessment was performed during the Week 20 visit.
Time Frame: Day -1 and Week 20: pre-infusion, post-infusion at multiple timepoints up to 96 hours
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Adynovate
Number analyzed (Participants) | 15
IU/dL
  Initial PK Assessment | 0 (0)
  Second PK Assessment: number analyzed (Participants) | 14
  Second PK Assessment | 0 (0)

29. Secondary Outcome: Terminal Phase Elimination Half-life (T1/2) for FVIII Activity Following an Initial Single Dose and Steady-state Dose of Adynovate
Description: T1/2 was calculated based on pre-infusion corrected concentration data. As per planned analysis, data for this outcome measure was collected and reported for initial PK assessment and second PK assessment. The initial PK assessment was performed prior to the baseline visit at Day -1. The second PK assessment was performed during the Week 20 visit.
Time Frame: Day -1 and Week 20: pre-infusion, post-infusion at multiple timepoints up to 96 hours
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Adynovate
Number analyzed (Participants) | 15
hour
  Initial PK Assessment | 16.0 (3.27)
  Second PK Assessment: number analyzed (Participants) | 14
  Second PK Assessment | 18.5 (4.61)

ADVERSE EVENTS:
Time Frame: Up to approximately 28 weeks
Description: The SAS included all participants treated with at least 1 Adynovate dose.
Groups:
- Adynovate: Participants received prophylactic treatment with Adynovate (45 [±5] IU/kg), infusion, IV, twice weekly, for at least 50 EDs or approximately 28 weeks.
Arm/Group | Adynovate
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 1/37
Other Adverse Events (participants affected / at risk) | 8/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adynovate (N=37)
Liver injury (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adynovate (N=37)
Alanine aminotransferase increased (Investigations) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Aspartate aminotransferase increased (Investigations) | 2
Diarrhoea (Gastrointestinal disorders) | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-04-16): https://cdn.clinicaltrials.gov/large-docs/51/NCT05707351/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT05707351/SAP_001.pdf